CLINICAL TRIAL: NCT00777179
Title: Randomized, Double-blinded, Placebo-controlled Phase II Study of Vandetanib (ZactimaTM) Maintenance for Locally Advanced or Metastatic Non-small-cell Lung Carcinoma (NSCLC) Following Platinum-doublet Chemotherapy
Brief Title: Phase II of Zactima Maintenance for Locally Advanced or Metastatic Non-small-cell Lung Carcinoma (NSCLC) Following Platinum-doublet Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4200C00077
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: NSCLC
Keywords: Vandetanib, NSCLC, Maintenance, Phase II
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vandetanib (Experimental)
  Interventions: Drug: Vandetanib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vandetanib — Tablet, oral, daily
  Other Names: Zactima TM
  Arms: Vandetanib
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is multicenter, randomized, double-blinded, placebo-controlled Phase II study comparing vandetanib (300mg daily) plus best supportive care (BSC) to placebo plus BSC as maintenance treatment in patients with locally advanced or metastatic NSCLC, who have received and responded to prior platinum-doublet systemic chemotherapy. The primary objective of the study is to compare the Progression Free Survival (PFS) rate at 3 months in locally advanced or metastatic NSCLC patients with or without vandetanib maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of locally advanced or metastatic NSCLC (IIIb-IV) at the time of original diagnosis.
* Completion of 4 cycles of chemotherapy of gemcitabine (1,000 or 1250mg/m^2/day on day 1 and 8) and cisplatin (70-80mg/m^2/day on day 1) every 3 weeks and have shown response, Complete Response(CR), Partial Response (PR) or stable disease (SD) by RECIST.
* WHO PS 0-1
* No prior radiotherapy to chest, immunotherapy or biologic therapy

Exclusion Criteria:

* Mixed small cell and non small-cell lung cancer history.
* Prior treatment with EGFR TKIs or VEGFR TKIs (prior treatment with cetuximab [Erbitux] or bevacizumab [Avastin] is not permitted.)
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol.
* Radiation therapy within 4 weeks before the start of study therapy. Major surgery within 4 weeks, or incomplete healed surgical incision before starting study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- South Korea (5):
  - Research Site, Cheongju-si, Republic of Korea
  - Research Site, Gyeonggi-do, Republic of Korea
  - Research Site, Gyeongsangnam-Do, Republic of Korea
  - Research Site, Incheon, Republic of Korea
  - Research Site, Seoul, Republic of Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 13 October 2008 Last patient enrolled: 7 December 2009 This study was conducted at Division of oncology, Department of Medicine of general hospitals in Korea.
Groups:
- Vandetanib: Vandetanib 300 mg, orally, once daily
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Vandetanib | Placebo
Started | 75 (Number of participants for intent-to-treat (ITT) set population) | 42 (Number of participants for intent-to-treat (ITT) set population)
Completed | 75 (All participants' data within ITT set were included for final result.) | 42 (All participants' data within ITT set were included for final result.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib | Placebo | Total
Number analyzed (Participants) | 75 | 42 | 117
Age, Customized [Median (Full Range); unit: year]
  Median (min-Max Range) | 61 [33 to 76] | 60.5 [29 to 70] | 61 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 14 | 42
  Male | 47 | 28 | 75
Smoking history [Number; unit: Participants]
  Smoker | 47 | 28 | 75
  Non-smoker | 28 | 14 | 42
Overall response at screening [Number; unit: Participants] — completion of 4 cycles of chemotherapy of gemcitabine (1,000mg/m^2/day or 1,250mg/m^2/day on day 1 and 8) and cisplatin (70mg/m^2/day~80mg/m^2/day on day 1) every 3 weeks and have shown responses (CR, PR) or stable disease (SD) by RECIST 1.0.
  Participants
    Partial Response (PR) | 44 | 30 | 74
    Stable Disease (SD) | 31 | 12 | 43
WHO Performance status [Number; unit: Participants] — WHO PS (0: Fully active, able to carry out all usual activities without restrictions and without the aid of analgesia. 1: Restricted in strenuous activity, but ambulatory and able to carry out light work or pursue a sedentary occupation. This group also contains subjects who are fully active, as in grade 0, but only with the aid of analgesics.)
  Participants
    0 | 20 | 10 | 30
    1 | 55 | 32 | 87
Histology [Number; unit: Participants] — Histology
  Participants
    Adenocarcinoma | 56 | 31 | 87
    Squamous cell carcinoma | 11 | 9 | 20
    Other | 8 | 2 | 10
Classification of lung tumor stage [Number; unit: Participants] — Classification (Stage IIIb: Any T - N3 - M0 or T4 - Any N - M0, Stage IV: Any T - Any N - M1)
  Participants
    Stage IIIb | 15 | 12 | 27
    Stage IV | 60 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate at 3 Months
Description: Progression-free survival (PFS) rate at 3 months is defined as the number of patients without evidence of progression or death after 3 months from randomisation among the PFS-evaluable patients.
Time Frame: 12 weeks
Population: The reported number of participants analyzed (Vandetanib: 63, Placebo: 38) are for PFS evaluable patient set.
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 63 | 38
Participants | 28 | 12

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) defined as the median time from randomization to death from any cause or first observed disease progression.
Time Frame: Performed at baseline, every 4 weeks until Week 12 following randomization and then every 8 weeks until objective disease progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 75 | 42
months | 2.7 [1.9 to 4.4] | 1.7 [0.9 to 2.6]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) defined as the median time from randomization to death from any cause.
Time Frame: Every 12 weeks unless the patient withdraws consent
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 75 | 42
months | 15.6 [9.6 to NA] — no maximum value, observation period for overall survival was not sufficient | 20.8 [15.2 to NA] — no maximum value, observation period for overall survival was not sufficient

4. Secondary Outcome: Disease of Response (DOR)
Description: Number of patients showing Complete Response (CR), Partial Response (PR) or Stable Disease (SD) based on RECIST for the best response.
  Number of patients showing Complete Response (CR, disappearance of all target lesions), Partial Response (PR, at least a 30% decrease in the sum of longest diameter of target lesions taking as reference the baseline sum longest diameter) or Stable Disease (SD, Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum longest diameter since the treatment started) based on RECIST Criteria Version 1.0 (assessed by CT and/or MRI) for the best response
Time Frame: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 75 | 42
Participants | 33 | 17

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Number of patients showing Complete Response (CR) or Partial Response (PR) based on RECIST for the best response.
  Number of patients showing Complete Response (CR, disappearance of all target lesions) or Partial Response (PR, at least a 30% decrease in the sum of longest diameter of target lesions taking as reference the baseline sum longest diameter) based on RECIST Criteria Version 1.0 (assessed by CT and/or MRI) for the best response.
Time Frame: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 75 | 42
Participants | 14 | 1

ADVERSE EVENTS:
Arm/Group | Vandetanib | Placebo
Serious Adverse Events (participants affected / at risk) | 18/75 | 4/42
Other Adverse Events (participants affected / at risk) | 72/75 | 37/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=75) | Placebo (N=42)
Pneumonia (Infections and infestations) | 12 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Transient ischemic attack (Nervous system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Convulsion (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Chest discomfort (Gastrointestinal disorders) | 2 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ileal perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=75) | Placebo (N=42)
Diarrhoea (Gastrointestinal disorders) | 45 | 4
Nausea (Gastrointestinal disorders) | 13 | 6
Anorexia (Metabolism and nutrition disorders) | 29 | 7
Insomnia (Psychiatric disorders) | 14 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 29 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 7
Constipation (Gastrointestinal disorders) | 8 | 2
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Stomatitis (Gastrointestinal disorders) | 8 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1
Asthenia (General disorders) | 9 | 3
Chest Discomfort (General disorders) | 7 | 2
Chest Pain (General disorders) | 12 | 5
Fatigue (General disorders) | 5 | 3
Mucosal Inflammation (General disorders) | 7 | 0
Pyrexia (General disorders) | 5 | 2
Hypersensitivity (Immune system disorders) | 0 | 5
Paronychia (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 9 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 4 | 3
Headache (Nervous system disorders) | 8 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 4
Anxiety (Nervous system disorders) | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Acne (Skin and subcutaneous tissue disorders) | 9 | 0
Flushing (Vascular disorders) | 6 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 10 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 58 | 11
Skin Lesion (Skin and subcutaneous tissue disorders) | 8 | 3
Hypertension (Vascular disorders) | 13 | 0
Vision blurred (Eye disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.